CLINICAL TRIAL: NCT06450977
Title: Remote Evaluation of MIND Diet
Acronym: REMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Naiman Khan, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REMIND
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis; Cognitive Change; Nutrition, Healthy
Keywords: Executive Function; MIND; Dietary Pattern; Telehealth
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIND Diet (Experimental): Participants in the active MIND diet group will be asked to consume one ready-to-eat meal per day from Daily Harvest® meal delivery service. The treatment meals will follow MIND diet guidelines and include leafy green vegetables, nuts, legumes, whole grains, berries, and extra virgin olive oil.
  Interventions: Other: MIND Diet
- Control Diet (Active Comparator): Participants in the control diet group will be asked to consume one ready-to-eat meal per day from Daily Harvest® meal delivery service. The Control group will receive daily meals that are isocaloric with the active/experimental meals but will follow a general diet based on the average American diet and Dietary Guidelines for Americans (i.e., vegetables, fruits, nuts, whole grains, and unsaturated fats).
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: MIND Diet — Daily meals designed to increase adherence to the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) dietary pattern.
  Arms: MIND Diet
Other: Control Diet — Daily meals designed to increase fruit, vegetable, and whole grain intake consistent with a healthy American diet.
  Arms: Control Diet

SUMMARY:
The goal of this clinical trial is to learn if increasing adherence to a Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet pattern improves thinking ability and memory compared to a healthy control diet in persons with Multiple Sclerosis (MS). The main question it aims to answer is:

Does the MIND diet improve cognitive performance relative to a control diet in persons with MS?

Participants will:

Consume one meal that follows the MIND diet or a control meal every day for 3 months, complete online surveys and cognitive testing before and after, and keep a record of the food they eat during the study.

DETAILED DESCRIPTION:
The purpose of this study is to understand how a healthy diet is related to thinking ability and memory in people with multiple sclerosis (MS). This study is fully remote consisting of meals being delivered to participant homes using Daily Harvest meal delivery service. Participants will be asked to consume a microwaveable study meal or prepackaged smoothie every day for 12 weeks. The study meals and smoothies will follow either a dietary pattern thought to improve brain health (Mediterranean-DASH Intervention for Neurodegenerative Delay; MIND), or a control diet, and will include foods commonly found in grocery stores. Participants will not know which diet they are assigned to (active or control). Participants will also be asked to follow simple dietary guidance on a healthy diet in addition to the meals provided. Participants will complete a series of online forms or surveys. Additionally, participants will complete an online cognitive battery from Cambridge Neuropsychological Test Automated Battery (CANTAB) at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18-64 years old
2. Self-reported diagnosis of Multiple sclerosis (MS)
3. 20/20 or corrected vision
4. No other neurodegenerative disease diagnosis
5. Stable disease-modifying therapy (DMT) within 6 months
6. Not Pregnant or lactating
7. No food allergies or intolerances
8. Able to consume study meals
9. Not enrolled in another dietary, exercise, or medication study during the study
10. Access to a computer/laptop with internet

Exclusion Criteria:

1. Individuals younger than 18 or older than 64 years old
2. No self-reported diagnosis of Multiple sclerosis (MS)
3. Not 20/20 or uncorrected vision
4. Other neurodegenerative disease diagnosis
5. Disease modifying therapy (DMT) less than 6 months
6. Pregnant or lactating
7. Food allergies or intolerances
8. Not able to consume study meals
9. Enrolled in another dietary, exercise, or medication study during the study
10. No access to a computer/laptop with internet

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Information Processing | 12 weeks (Baseline vs. Follow Up)
  Rapid Visual Information Processing Task from CANTAB online battery
Visual Processing | 12 weeks (Baseline vs. Follow Up)
  Match to Sample Visual Search from CANTAB online battery
Processing Speed | 12 weeks (Baseline vs. Follow Up)
  Digit Span from CANTAB online battery
Learning | 12 weeks (Baseline vs. Follow Up)
  Paired Associates Learning Task from CANTAB online battery
Memory | 12 weeks (Baseline vs. Follow Up)
  Spatial Working Memory from CANTAB online battery
MIND Scores | 12 weeks (Baseline vs. Follow Up)
  MIND dietary pattern scores calculated from diet records/surveys. Validated score to determine how someone adheres to the dietary pattern, scale of 0 to 14 with a higher score indicating greater adherence to the pattern.

SECONDARY OUTCOMES:
Recruitment Rates | Throughout the recruitment process
  Measure the number of participants contacted and interested in participating in the study
Refusal Rates | Throughout the recruitment process.
  Measure the number of participants that refused to participate in the intervention. Data on refusal factors will be collected through emails and calls and summarized.
Retention rates | Throughout the intervention (weeks 1-12)
  Retention will be described as the proportion of enrolled participants who complete the intervention
Attrition rates | Throughout the intervention (weeks 1-12)
  Attrition is the proportion of the participants who did not complete the intervention.
Adherence/Compliance Rates | Throughout the intervention (weeks 1-12)
  Adherence rates are the proportion of intervention meals and guidelines the participants followed. These will be tracked through tracking surveys throughout the intervention.
Participant Experience and Burden | Throughout the intervention (weeks 1-12)
  Participants will report feedback on the intervention through video chats. Descriptives of participant experience and burden of intervention will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Naiman Khan, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No